CLINICAL TRIAL: NCT01693328
Title: A French, Multicentre, Open-label, Observational Study to Assess Quality of Life and Satisfaction in Subjects Taking PecFent® for the Treatment of Breakthrough Cancer Pain (BTPc)
Brief Title: Patient Satisfaction and Quality of Life Impact - PecFent®
Acronym: Qualipec
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Archimedes Development Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CP057/11
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Breakthrough Cancer Pain
Keywords: quality of life; PecFent; Lazanda; fentanyl; intranasal; breakthrough cancer pain
MeSH Terms: interventions — Fentanyl; Nasal Sprays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PecFent®
  Interventions: Drug: PecFent® (fentanyl) nasal spray

INTERVENTIONS:
Drug: PecFent® (fentanyl) nasal spray

SUMMARY:
National multicenter, prospective, observational study in cancer patients with chronic background pain and breakthrough pain to whom PecFent® has been prescribed under pragmatic condition by a specialist in the treatment of cancer pain conditions.

• Study objectives include assessment of early treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged ≥18 years) with cancer
* Taking at least 60 mg of oral morphine sulfate or equivalent per day for chronic background pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with breakthrough pain
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Satisfaction | Satisfaction will be assessed approximately 1 hour after each BTPc episode treated with PecFent® from completion of titration through Day 7
  Satisfaction will be assessed using a 4-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Serrie, MD, Principal Investigator — Head of Pain Federation - Palliative Medicine Lariboisiere Hospital, Paris France
Locations (1):
- Centre Léon-Bérard, Lyon, France